CLINICAL TRIAL: NCT05465239
Title: Intelligent and Adaptive Control Applied to Powered Walkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of Virginia (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SurePace1; 2R44HD082863-02 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SurePace Powered Walker User (Experimental): Before any formal experiments are conducted, participants will be given an opportunity to "train" with the new powered walker for a pre-defined period of time to eliminate the confounding effects of being unfamiliar with using the device. (See the description of UVA's facilities and Protection of Human Subjects document for additional discussion of safety measures/protocols and Institutional Review Board procedures.) Experiments will consist of one-hour sessions (with adequate rest periods between trials and time for evaluations) in which participants will be asked to walk at a self-selected (comfortable) walking speed through a pre-defined 8 m x 4 m oval course.
  Interventions: Device: SurePace Powered Walker User

INTERVENTIONS:
Device: SurePace Powered Walker User — Participants will be asked to perform one baseline 5-minute trial with the lab's instrumented walker in passive mode (no powered locomotion) and two 5-minute trials with the walker in active mode (powered locomotion).

SUMMARY:
The research is towards an advanced control and computer learning strategy that will intelligently drive a powered walker for people with walking disabilities. The aim of the control strategy is to provide powered assistance that optimally reduces the metabolic cost of walking. The goal of the proposed intelligent walker is to reduce the workload of walking, keeping this population walking longer, providing critical exercise, continued muscle development and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

Typically developed subjects:

• No walking disabilities

Subjects with CP:

* Diagnosed with spastic CP
* GMFCS level II-III
* Ages 5-25 inclusive
* No surgeries in last 6 months
* Able to ambulate 40ft unaided (excluding walker)
* Understand and follow commands

Exclusion Criteria:

Typically developed subjects:

• Observed intramuscular pathology

Subjects with CP:

* Mental retardation
* Severe uncontrolled seizures
* Leg or foot surgery in last 12 months
* Surgery or significant injury in last 6 months affecting
* walking ability
* Inability to ambulate unassisted (other than walker) 40ft
* without stopping to rest
* Inability to understand or follow commands

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Burkholder, Ph.D., Principal Investigator — Barron Associates, Inc.
Locations (1):
- University of Virginia Motion Analysis and Motor Performance Lab, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at the University of Virginia medical center. The first participant was enrolled in December 2020 and the last participant was enrolled in September 2023.
Pre-assignment Details: 48 enrolled participants met the inclusion criteria and completed the study.
Groups:
- Control Subjects: Before any formal experiments are conducted, participants will be given an opportunity to "train" with the new powered walker for a pre-defined period of time to eliminate the confounding effects of being unfamiliar with using the device. (See the description of UVA's facilities and Protection of Human Subjects document for additional discussion of safety measures/protocols and Institutional Review Board procedures.) Experiments will consist of one-hour sessions (with adequate rest periods between trials and time for evaluations) in which participants will be asked to walk at a self-selected (comfortable) walking speed through a pre-defined 8 m x 4 m oval course.
  SurePace Powered Walker User: Participants will be asked to perform one baseline 5-minute trial with the lab's instrumented walker in passive mode (no powered locomotion) and two 5-minute trials with the walker in active mode (powered locomotion).
- Walking Disability Subjects: Subjects with walking disabilities, such as cerebral palsy (CP). Before any formal experiments are conducted, participants will be given an opportunity to "train" with the new powered walker for a pre-defined period of time to eliminate the confounding effects of being unfamiliar with using the device. (See the description of UVA's facilities and Protection of Human Subjects document for additional discussion of safety measures/protocols and Institutional Review Board procedures.) Experiments will consist of one-hour sessions (with adequate rest periods between trials and time for evaluations) in which participants will be asked to walk at a self-selected (comfortable) walking speed through a pre-defined 8 m x 4 m oval course.
  SurePace Powered Walker User: Participants will be asked to perform one baseline 5-minute trial with the lab's instrumented walker in passive mode (no powered locomotion) and two 5-minute trials with the walker in active mode (powered locomotion).
Period: Overall Study
Arm/Group | Control Subjects | Walking Disability Subjects
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Subjects: Normally developed subjects without walking disabilities.
- Walking Disability Subjects: Subjects with walking disabilities, such as cerebral palsy.
- Total: Total of all reporting groups
Arm/Group | Control Subjects | Walking Disability Subjects | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (17.2) | 15.5 (5.6) | 15.8 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 9 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 3 | 4
  White | 21 | 17 | 38
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Cost (Oxygen Consumption)
Description: Oxygen consumption data will be collected with a Oxycon Mobile (VIASYS Healthcare Inc.) portable indirect calorimetry system. The outcome measure is the reduction in metabolic cost of using the powered walker compared to an unpowered walker.
Time Frame: Five minutes
Measure: Mean (Standard Deviation); unit: J/kg
Groups:
- Control Subjects: Unpowered Walker: Normally developed subjects without walking disabilities.
- Walking Disability Subjects: Unpowered Walker: Subjects with walking disabilities, such as cerebral palsy.
- Control Subjects: Powered Walker: Normally developed subjects using Powered Walker
- Walking Disability Subjects: Powered Walker: Subjects with walking disabilities, such as cerebral palsy, using the powered walker.
Arm/Group | Control Subjects: Unpowered Walker | Walking Disability Subjects: Unpowered Walker | Control Subjects: Powered Walker | Walking Disability Subjects: Powered Walker
Number analyzed (Participants) | 24 | 24 | 24 | 24
J/kg | 11.0 (2.9) | 12.7 (3.3) | 7.0 (1.2) | 9.4 (3.5)
Statistical Analysis 1: Comparison: Control Subjects: Unpowered Walker vs Control Subjects: Powered Walker; Test type: Equivalence — Equivalence analysis of metabolic energy consumption using the unpowered vs powered walker for control subjects; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Walking Disability Subjects: Unpowered Walker vs Walking Disability Subjects: Powered Walker; Test type: Equivalence — Equivalence analysis of metabolic energy consumption using the unpowered vs powered walker for subjects with walking disabilities; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Through study completion, which was a single session, an average of 2 hours.
Groups:
- Control Subjects: Unpowered Walker: Normally developed subjects without walking disabilities using unpowered walker.
- Walking Disability Subjects: Unpowered Walker: Subjects with walking disabilities, such as cerebral palsy, using unpowered walker.
- Control Subjects: Powered Walker: Normally developed subjects without walking disabilities using powered walker.
- Walking Disability Subjects: Powered Walker: Subjects with walking disabilities, such as cerebral palsy, using powered walker.
Arm/Group | Control Subjects: Unpowered Walker | Walking Disability Subjects: Unpowered Walker | Control Subjects: Powered Walker | Walking Disability Subjects: Powered Walker
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05465239/Prot_SAP_000.pdf